CLINICAL TRIAL: NCT04539353
Title: The Association Between Pain Intensity and Heart Rate Variability in Chronic Pain Patients.
Brief Title: HRV and Pain Intensity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Moens Maarten (Other)
Responsible Party: Sponsor-Investigator, Moens Maarten, principal investigator, Universitair Ziekenhuis Brussel
Organization: Universitair Ziekenhuis Brussel (Other)
Other Study IDs: INTERVAL
Record Dates: First submitted 2020-08-26; First posted 2020-09-07 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- chronic pain: Patients with chronic pain, regardless of the cause of the pain.
  Interventions: Other: Heart Rate Variability; Other: Pain intensity

INTERVENTIONS:
Other: Heart Rate Variability — Heart Rate Variability will be measured with a Polar device.
Other: Pain intensity — Pain Intensity will be measured with a Numeric Rating Scale and Visual Analogue Scale

SUMMARY:
The aim of this study is to explore the association between pain intensity and heart rate variability in patients with chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic pain for at least 3 months
* Age > 18 years
* Patient has been informed of the study procedures and has given written informed consent
* Patient willing to comply with study protocol

Exclusion Criteria:

* Healthy patients or patients with acute pain.
* Evidence of an active disruptive psychiatric disorder that may impact perception of pain, and/or ability to evaluate treatment outcome as determined by investigator
* Patients were excluded if they had one or more coexisting conditions known to affect HRV analysis.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Chronic pain patients (regardless of the cause of the pain).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-12-14 (Actual); Primary Completion 2021-10-15 (Estimated); Study Completion 2021-10-15 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Variability | During study visit, cross-sectional, once, during 5 minutes.
  Heart Rate Variability will be measured with a Polar device during a 5 minute recording.
Pain Intensity with Numeric Rating Scale | During study visit, cross-sectional, once.
  Pain Intensity will be measured with a Numeric Rating Scale.
Pain Intensity with Visual Analogue Scale | During study visit, cross-sectional, once.
  Pain Intensity will be measured with a Visual Analogue Scale.

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Universitair Ziekenhuis Brussel, Jette
  - AZ Delta, Roeselare

REFERENCES:
- [Derived] Moens M, Billet B, Molenberghs G, De Smedt A, Pilitsis JG, De Vos R, Hanssens K, Billot M, Roulaud M, Rigoard P, Goudman L. Heart rate variability is not suitable as a surrogate marker for pain intensity in patients with chronic pain. Pain. 2023 Aug 1;164(8):1741-1749. doi: 10.1097/j.pain.0000000000002868. Epub 2023 Jan 19. PMID 36722463